CLINICAL TRIAL: NCT02031315
Title: Sudden Death in Sub-Saharan Africa: Design and Protocol of The DOUALA-SD Prospective Survey
Brief Title: Epidemiology of Sudden Death in Cameroon
Acronym: DOUALA-SD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cameroon Resuscitation Council (Other)
Collaborators: ARCV (Unknown)
Responsible Party: Principal Investigator, BONNY Aimé, Chief manager, Cameroon Resuscitation Council
Other Study IDs: CRC-SD 2013
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Diseases
Keywords: sudden death; sudden cardiac arrest
MeSH Terms: conditions — Cardiovascular Diseases; Death, Sudden; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 72 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Resident of health areas of interest: Residents of 4 health areas will be monitored for sudden unexpected death within 72 months of follow up. Circumstances and past medical conditions will be checked.

SUMMARY:
Background The burden of sudden death (SD) in sub-Saharan Africa is unknown. The aim is to assess the incidence, etiology and patient characteristics of SD in a sub-Saharan country. Methods The Douala-SD study is a prospective, multicenter, community-based registry monitoring all cases of SD occurring in index areas of Douala city. Investigators will use the definition of SD as natural death occurring within 24h at the onset of symptoms. Demographic, clinical, electrocardiographic and biological variables (when available) of victims will be recorded. All deaths occurring in residents of health areas of interest will be checked for past medical history, circumstances of death, and autopsy (if possible). Conclusion This maiden Douala-SD study will provide comprehensive, contemporary data on the epidemiology of SD in a sub-Saharan African country and will help in the development of strategies to prevent and manage SD in Africa.

DETAILED DESCRIPTION:
Two health areas were excluded for inaccurate data collection, and 2 other were randomly disqualified as investigators previously decided to conduct the survey in ≤ 4 areas. The mode of randomization aimed at includes no more than 1 health area per district. Finally, investigators retained 4 health areas representing 4 out of 6 districts of Douala. Thus, the sampling of 240,384 inhabitants will be monitored prospectively. All administrative staff and community-healthcare committee, the so-called " comité de santé" (COSA) of each health area will be a key component of the research team, helping identify every case of death in the area of concern. Every case of death will be reported by the staff of COSA in a specific questionnaire form. In addition to the deaths noted by members of each COSA, investigators will pay attention with all notices of deaths in local newspapers, radio, interrogation of health area residents, and death certificates from local medical centers.

ELIGIBILITY:
Inclusion Criteria: All witnessed and unwitnessed victims of unexpected natural death

-

Exclusion Criteria:

* Victims living in the area of interest for a short time frame (< 12 months)
* Absence of information helping to determine circumstances of death

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: First, the subject must be a permanent resident of one of 4 'health areas' included in the study. Second, each district of interest must have an updated population census.
Sampling Method: Probability Sample
Enrollment: 240000 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Sudden death, either cardiac or non-cardiac origin | one year

CONTACTS AND LOCATIONS:
Overall Officials: Aimé BONNY, MD, Principal Investigator — Teaching Hospital Laquintinie, University of Douala, Cameroon
Locations (1):
- Cameroon Resuscitation Council, Douala, Cameroon

REFERENCES:
- [Background] Arthur JT. Sudden deaths: cardiac and non-cardiac in children in Accra. West Afr J Med. 1995 Apr-Jun;14(2):108-11. PMID 7495711
- [Background] Akinwusi PO, Komolafe AO, Olayemi OO, Adeomi AA. Pattern of sudden death at Ladoke Akintola University of Technology Teaching Hospital, Osogbo, South West Nigeria. Vasc Health Risk Manag. 2013;9:333-9. doi: 10.2147/VHRM.S44923. Epub 2013 Jun 24. PMID 23836978